CLINICAL TRIAL: NCT00576641
Title: A Phase l Trial of Tumor Associated Antigen Pulsed Dendritic Cell Immunotherapy for Patients With Brain Stem Glioma and Glioblastoma
Brief Title: Immunotherapy for Patients With Brain Stem Glioma and Glioblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Surasak Phuphanich, MD, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6657
Record Dates: First submitted 2007-12-18; First posted 2007-12-19 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2014-10

CONDITIONS: Brain Stem Glioma; Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vaccine (Experimental)
  Interventions: Biological: autologous dendritic cells

INTERVENTIONS:
Biological: autologous dendritic cells

SUMMARY:
The purpose of the Dendritic Cell Immunotherapy study for patients with glioblastoma and/or brainstem glioma is to determine whether in patients with malignant brain tumors, dendritic cells injected peripherally can reactivate the immune system against the brain tumor.

DETAILED DESCRIPTION:
Patients will have their white blood cells removed and grown in culture under conditions to make dendritic cells. Dendritic cells are a small group of cells that belong to the white blood cell population. These cells are responsible for letting the immune system know that something foreign, like bacteria or a tumor, is in the body. Dendritic cells help the body ward off disease by alerting the immune system. In previous clinical trials, brain tumor cells called astrocytoma tumor cells and glioblastoma tumor cells were taken from the tumor that was removed during surgery. The brain tumor cells were then placed into a solution in the laboratory that made them grow. Certain parts of the brain tumor's proteins (peptides) were removed from the growing tumor cells and mixed together with the dendritic cells in the blood taken from a vein. This combination of dendritic cells and brain tumor peptides were injected into the patient's skin, like a vaccination. This process is similar to that used in vaccinations. The patients were given three and four injections of dendritic cells mixed with the tumor peptides over the course of a twenty-eight day period.

In this study, the proteins that are manufactured and known to be associated with brain cancers will be mixed with the dendritic cells obtained during leukopheresis (a procedure in which the dendritic cells are separated from the patients' blood). They will then undergo three vaccinations along with follow up clinic visits (which include evaluations and laboratory tests) to check their status.

The investigators learned that it was possible to generate an immune response in a subset of patients with malignant glioma. In addition, these cells were able to reach the brain and kill brain tumor cells. The survival of patients in this study was prolonged when compared to historical controls. Based on clinical data in subjects with brain tumors, the investigators believe that peripheral injection of dendritic cells will generate a more potent immune response for patients with brain stem gliomas and/or glioblastomas. The investigators hope to determine whether this therapy will translate into a longer survival and better quality of life in these patients in whom survival is measured in months. Through this study the investigators hope to learn more about the role of the body's immune response against cancer and about the use of dendritic cells for immunotherapy. This information may prove useful in the therapy of patients with glioblastoma and/or brainstem gliomas.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be HLA -A1 or HLA - A2 positive
* Both male and female of child bearing age must use medically accepted form of birth control
* Confirmed brain stem glioma and glioblastoma with MRI
* Presence of at least one of the antigens by immunohistochemistry
* Karnofsky performance of at least 60%
* On maintenance glucocorticoid therapy at no more 2 mg BID
* Hematologic and chemistry profiles within the parameters of the protocol
* Wash ou periods from previous therapies: 6 weeks from nitrosurea, 4 weeks from chemotherapy, 2 weeks after resolution of Grade 3 or 4 toxicity
* Able to sign IRB approved Informed consent
* Three adults will be treated prior to any study agent administration to subjects younger than 18 years of age

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2007-05; Primary Completion 2010-01 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Evaluate safety/toxicity of Dendritic cell vaccine, Monitor survival and time to progression and monitor the cellular immune responses. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Surasak Phuphanich, M.D., Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Jouanneau E, Black KL, Veiga L, Cordner R, Goverdhana S, Zhai Y, Zhang XX, Panwar A, Mardiros A, Wang H, Gragg A, Zandian M, Irvin DK, Wheeler CJ. Intrinsically de-sialylated CD103(+) CD8 T cells mediate beneficial anti-glioma immune responses. Cancer Immunol Immunother. 2014 Sep;63(9):911-24. doi: 10.1007/s00262-014-1559-2. Epub 2014 Jun 4. PMID 24893855